CLINICAL TRIAL: NCT03217513
Title: Pilot Study to Evaluate Knee Osteoarthritis Outcome Measures in Arthritic Patients Prescribed Forteo or Prolia for Osteoporosis
Brief Title: Knee Osteoarthritis Outcome Measures in Arthritic Patients With Osteoporosis
Status: Withdrawn | Type: Observational
Why Stopped: never started
Sponsor: Edward Fox (Other)
Responsible Party: Sponsor-Investigator, Edward Fox, Principal Investigator/Sponsor, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Other Study IDs: STUDY00004918
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Osteoporosis; Knee Osteoarthritis
Keywords: osteoporosis; osteoarthritis; knee
MeSH Terms: conditions — Osteoporosis; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Forteo: teriparatide 20-microgram once daily available in a 2.4-mL delivery device for subcutaneous injection by the patient
- Prolia: denosumab 60 mg administered as a single subcutaneous injection every 6 months by the health care provider

SUMMARY:
The purpose of this study is to generate proof of concept human data by evaluating osteoarthritis outcome measures in arthritic patients that are prescribed Forteo® as the standard of care to treat their primary diagnosis of osteoporosis.

DETAILED DESCRIPTION:
The traditional treatment paradigm for osteoarthritis (OA) involves palliative strategies focused on pain management and joint replacement. The longstanding inability to develop disease-modifying therapies that can rejuvenate joint cartilage is a great unmet need considering that diarthrodial and spinal OA is the most prevalent disease in the US, equal in numbers to the next top 4 disorders combined (heart, pulmonary, mental health and diabetic conditions) (CDC, 2009). Thus, the development of an effective remittive treatment for OA is a vital public health initiative with potential for tremendous impact. Our long-term research objective is to test a radically different strategy for treatment of OA that is based on findings recently published in Science Translational Medicine (Sampson et al., 2011) that identified human parathyroid hormone1-34 (teriparatide) as a chondroregenerative agent in a murine model of OA. Suggesting a parallel effect in human OA, data mined from the NIH-sponsored OA Initiative revealed improved WOMAC knee function scores in arthritic subjects coincidentally prescribed teriparatide (trade name: Forteo®) to treat osteoporosis. These preclinical and human data provide compelling rationale to study Forteo® as a novel OA therapy directed at improving joint structure and function. The central aim of our overall research program is to challenge the paradigm that cartilage loss in OA is irreversible. Thus, our long-term programmatic goal is to test Forteo® as the first and only disease-modifying treatment for OA with potential to rapidly impact clinical care. To achieve this, we have been developing a clinical trial where subjects with medial compartment Kellgren Lawrence (K-L) stage II-III knee OA will receive either Forteo® or Prolia® (a brand of denosumab) for two years. Disease progression will be assessed via structural, biomarker and functional outcomes at various time points out to 24 months post-initiation of therapy. Since Forteo® is a widely used therapeutic in patients with osteoporosis (OP)-related severe bone loss, we propose to examine OA outcomes in OP patients with concomitant knee OA. This pilot study described here that tests the hypothesis that patients with unilateral or bilateral knee OA (Kellgren-Lawrence grade II-III) that are prescribed Forteo® to treat their primary diagnosis of OP will demonstrate improved physical function (Timed-Up-And-Go), improved patient-reported outcomes (PROMIS 12a, v1.0), and increased blood levels in the cartilage anabolic marker type II collagen C-propeptide. Completion of this proposed experimental design would provide critical proof-of-concept preliminary data supporting the use of biomarkers, physical function testing and questionnaire-based functional assessment to study OA in patients.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age: 40-80 years (inclusive)
* Gender: male or female (non-pregnant)
* Fluent in written and spoken English
* Patients capable of giving informed consent
* Primary diagnosis of osteoporosis that will be treated with either Forteo® to induce bone anabolism or Prolia® by the study investigator as part of patient's standard of care treatment
* Symptomatic, medial compartment knee OA with a Kellgren-Lawrence (K-L) score between II-III (documented in the medical record by previously collected knee series radiography). Radiographs to be performed within past two years.

EXCLUSION CRITERIA:

* Age < 40 or >80 years
* Cognitive impairment
* Pregnancy
* Non-English speaking persons
* History of hyperparathyroidism, hypercalcemia, current/recent renal stones, or malignancy
* Depression (currently taking home medication)
* History of inflammatory disease (colitis, rheumatoid arthritis, psoriasis, lupus, scleroderma, spondylitis)
* Use of immunosuppressants, chemotherapy, or radiotherapy
* BMI, angular deformity and K-L score of the contralateral knee (if the OA is bilateral) will be noted as covariates

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that are evaluated, treated, and followed by the study investigator
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood levels | 2 years
  Type II collagen degradation neoepitope and C-propeptide

SECONDARY OUTCOMES:
Urine levels | 2 years
  Type II collagen C-telopeptide
Physical function | 2 years
  Timed-Up-And-Go
Patient reported outcomes | 2 years
  PROMIS SF v1.0-Physical Function 12a

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Fox, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aletaha D. From the item to the outcome: the promising prospects of PROMIS. Arthritis Res Ther. 2010;12(1):104. doi: 10.1186/ar2910. Epub 2010 Feb 1. PMID 20156319
- [Background] Bischoff-Ferrari HA, Vondechend M, Bellamy N, Theiler R. Validation and patient acceptance of a computer touch screen version of the WOMAC 3.1 osteoarthritis index. Ann Rheum Dis. 2005 Jan;64(1):80-4. doi: 10.1136/ard.2003.019307. Epub 2004 Jul 1. PMID 15231508
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence and most common causes of disability among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2009 May 1;58(16):421-6. PMID 19407734
- [Background] Fries JF, Krishnan E, Rose M, Lingala B, Bruce B. Improved responsiveness and reduced sample size requirements of PROMIS physical function scales with item response theory. Arthritis Res Ther. 2011;13(5):R147. doi: 10.1186/ar3461. Epub 2011 Sep 14. PMID 21914216
- [Background] Sampson ER, Hilton MJ, Tian Y, Chen D, Schwarz EM, Mooney RA, Bukata SV, O'Keefe RJ, Awad H, Puzas JE, Rosier RN, Zuscik MJ. Teriparatide as a chondroregenerative therapy for injury-induced osteoarthritis. Sci Transl Med. 2011 Sep 21;3(101):101ra93. doi: 10.1126/scitranslmed.3002214. PMID 21937758
- [Background] Brostrom EW, Esbjornsson AC, von Heideken J, Iversen MD. Gait deviations in individuals with inflammatory joint diseases and osteoarthritis and the usage of three-dimensional gait analysis. Best Pract Res Clin Rheumatol. 2012 Jun;26(3):409-22. doi: 10.1016/j.berh.2012.05.007. PMID 22867935
- [Background] Kraus VB, Feng S, Wang S, White S, Ainslie M, Brett A, Holmes A, Charles HC. Trabecular morphometry by fractal signature analysis is a novel marker of osteoarthritis progression. Arthritis Rheum. 2009 Dec;60(12):3711-22. doi: 10.1002/art.25012. PMID 19950282
- [Background] Garnero P, Thompson E, Woodworth T, Smolen JS. Rapid and sustained improvement in bone and cartilage turnover markers with the anti-interleukin-6 receptor inhibitor tocilizumab plus methotrexate in rheumatoid arthritis patients with an inadequate response to methotrexate: results from a substudy of the multicenter double-blind, placebo-controlled trial of tocilizumab in inadequate responders to methotrexate alone. Arthritis Rheum. 2010 Jan;62(1):33-43. doi: 10.1002/art.25053. PMID 20039425
- [Background] Hashimoto J, Garnero P, van der Heijde D, Miyasaka N, Yamamoto K, Kawai S, Takeuchi T, Yoshikawa H, Nishimoto N. A combination of biochemical markers of cartilage and bone turnover, radiographic damage and body mass index to predict the progression of joint destruction in patients with rheumatoid arthritis treated with disease-modifying anti-rheumatic drugs. Mod Rheumatol. 2009;19(3):273-82. doi: 10.1007/s10165-009-0170-4. Epub 2009 May 19. PMID 19452245
- [Background] Maksymowych WP, Poole AR, Hiebert L, Webb A, Ionescu M, Lobanok T, King L, Davis JC Jr. Etanercept exerts beneficial effects on articular cartilage biomarkers of degradation and turnover in patients with ankylosing spondylitis. J Rheumatol. 2005 Oct;32(10):1911-7. PMID 16206346
- [Background] Papuga MO, Beck CA, Kates SL, Schwarz EM, Maloney MD. Validation of GAITRite and PROMIS as high-throughput physical function outcome measures following ACL reconstruction. J Orthop Res. 2014 Jun;32(6):793-801. doi: 10.1002/jor.22591. Epub 2014 Feb 14. PMID 24532421
- [Background] Taylor ME, Delbaere K, Mikolaizak AS, Lord SR, Close JC. Gait parameter risk factors for falls under simple and dual task conditions in cognitively impaired older people. Gait Posture. 2013 Jan;37(1):126-30. doi: 10.1016/j.gaitpost.2012.06.024. Epub 2012 Jul 23. PMID 22832468
- [Background] Debi R, Mor A, Segal G, Segal O, Agar G, Debbi E, Halperin N, Haim A, Elbaz A. Correlation between single limb support phase and self-evaluation questionnaires in knee osteoarthritis populations. Disabil Rehabil. 2011;33(13-14):1103-9. doi: 10.3109/09638288.2010.520805. Epub 2011 Jan 5. PMID 21208029